CLINICAL TRIAL: NCT00444483
Title: Structured Treatment and Teaching of Elderly Patients With Type 2 Diabetes Mellitus
Brief Title: Structured Patient Education and Quality of Life of Elderly Patients With Diabetes Mellitus- a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: University of Jena (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0099-9/98 (KIMII)-955
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Impact of Structured DTTP on Quality of Life; Insulin Therapy; Metabolic Control; Psychological Aspects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Structured diabetes teaching and treatment program

SUMMARY:
The improvement of the quality of life (QoL) is one of the key treatment goals in patients with diabetes mellitus. Objective: Prospective study to evaluate the impact of structured diabetes education on the QoL in insulin-treated, elderly patients with type 2 diabetes mellitus. Inpatients with insulin treated type 2 diabetes or failure of oral antidiabetic therapy were successively recruited and participated in the structured inpatient diabetes treatment and teaching program (DTTP) for insulin therapy QoL was assessed before and six months after participation in the DTTP with the standardised questionnaire of Lohr analysing the subscales: social relations, physical complaints, worries about the future, diet restrictions, fear of hypoglycemia, and daily struggles.

DETAILED DESCRIPTION:
All patients with type 2 diabetes mellitus, who were older than 54 years and admitted by general practitioner to the inpatient unit of the university hospital of Jena, Germany, for participation in a structured DTTP for insulin therapy because of hyperglycemia, were candidates for successive inclusion in the study. All patients participated in a five day inpatient structured DTTP for single or split dose administration of intermediate-acting insulin which included instruction in insulin injection, self- monitoring, hypoglycemia, acute/late complications, nutrition and foot care. Quality of life was assessed by using a validated instrument, the standardised QoL- questionnaire of Lohr et al. (21) both before and six months after participation in the DTTP. This questionnaire consists of 58 Likert- scaled items comprising the subscales: social relations, physical complaints, worries about the future, diet restrictions, fear of hypoglycemia, and daily struggles. Higher scores reflect higher quality of life with 100% as an optimum quality of life. The primary outcome measure regarding patients metabolic control was the improvement of quality of life six months after DTTP.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus, insulin therapy, age >54 years, hyperglycemia

Exclusion Criteria:

* dementia, severe neurological deficits, polioencephalitis, rejection of informed consent

Min Age: 54 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50

PRIMARY OUTCOMES:
The primary outcome measure regarding patients metabolic control was the improvement of quality of life six months after DTTP.

SECONDARY OUTCOMES:
A secondary objective of the study was the comparison of QoL- subscale in patients already on insulin therapy with those newly on insulin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Müller, MD, Principal Investigator — University of Jena; Anke Braun, MD, Study Chair — Bethanien Hospital Heidelberg, Germany; Ralf Schiel, MD, Study Chair — Inselklinik Heringsdorf, Germany